CLINICAL TRIAL: NCT06665516
Title: Frequency and Impact of Iron Deficiency in Pain Clinic Patients
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Other Study IDs: BRID
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2024-10

CONDITIONS: Iron Deficiency; Fibromyalgia
Keywords: iron deficiency; fibromyalgia; iron infusion therapy; chronic pain; pain management; diet; sex and gender; women's health; serotonin
MeSH Terms: conditions — Iron Deficiencies; Fibromyalgia; Chronic Pain; Agnosia; Coitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to measure the proportion of patients who have iron deficiency and if iron deficiency is treated what is the outcome. Participants will fill out a questionnaire to assess positive impact of iron supplementation treatment to assess whether they are at potential risk of iron deficiency

DETAILED DESCRIPTION:
The study is an observational clinical audit, with an unblinded clinical intervention. Iron deficiency and some chronic pain syndromes like fibromyalgia are more common in women of reproductive age. Iron deficiency can present with symptoms that are similar to those of fibromyalgia, but once recognized, iron deficiency is typically easily treated. The investigators intend to poll patients at the DeGroote Pain Clinic based on information from studies conducted in Australia and Great Britain. The investigators will determine who is at risk for iron deficiency based upon symptoms such as heavy periods, history of pregnancy, blood donation, diet, and any previous iron deficiency. The investigators will then confirm the results with lab testing, and provide treatment if necessary. The goal is to find out the percentage of women with chronic pain who also have iron deficiency, and assess the effect of treating iron deficiency on their pain symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patient at the DeGroote Pain Clinic
* Menstruating women between the ages of 18-49
* Willingness to complete the questionnaire, and undergo laboratory tests if indicated.

Exclusion Criteria:

* The only exclusion criteria is unwillingness to participate

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Cisgender women
Study Population: Female patients attending the DeGroote Pain Clinic
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-06-09 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients at risk of iron deficiency at the DeGroote Pain Clinic | from enrollment to end of treatment after 3 months
  Our primary outcome is the proportion of the 81 patients who are at risk of iron deficiency. This will be measured through positive questionnaire responses with symptoms/conditions that indicate risk of iron deficiency. Women patients arriving for pain clinic visits will be asked if they wish to participate in this audit and complete a screening questionnaire.The questionnaire determines high risk for Iron Deficiency through known risk factors: heavy menstrual bleeding, previous iron status, and iron supplementation. Previous studies identified heavy menstrual bleeding as a significant predictor of anemia and progression into ID.7 Patients were asked to report any of the four major symptoms (need double sanitary protection, need to frequently change your protection, had or worried about flooding through to clothes or bedding, pass large blood clots.), with a yes to 2 or more being considered to describe heavy menstrual bleeding and therefore high risk for experiencing iron deficiency.

CONTACTS AND LOCATIONS:
Locations (1):
- DeGroote Pain Clinic, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
IPD is not planned to be shared as this is a pilot study analysing the feasability of treatment. If successful, this can be scaled up nationwide at which point IPD will be shared.

REFERENCES:
- [Result] Murray CJL; GBD 2021 Collaborators. Findings from the Global Burden of Disease Study 2021. Lancet. 2024 May 18;403(10440):2259-2262. doi: 10.1016/S0140-6736(24)00769-4. No abstract available. PMID 38762327
- [Result] GBD 2021 Anaemia Collaborators. Prevalence, years lived with disability, and trends in anaemia burden by severity and cause, 1990-2021: findings from the Global Burden of Disease Study 2021. Lancet Haematol. 2023 Sep;10(9):e713-e734. doi: 10.1016/S2352-3026(23)00160-6. Epub 2023 Jul 31. PMID 37536353
- [Result] Pasricha SR, Tye-Din J, Muckenthaler MU, Swinkels DW. Iron deficiency. Lancet. 2021 Jan 16;397(10270):233-248. doi: 10.1016/S0140-6736(20)32594-0. Epub 2020 Dec 4. PMID 33285139
- [Result] Dugan C, MacLean B, Cabolis K, Abeysiri S, Khong A, Sajic M, Richards T; Women's Health research Collaborative. The misogyny of iron deficiency. Anaesthesia. 2021 Apr;76 Suppl 4:56-62. doi: 10.1111/anae.15432. PMID 33682094
- See also: This website provides a clear and concise summary of the information we will be investigating in this trial. This was provided to us by Dr. Toby Richards, the author of the website — https://www.theironclinic.com/iron-treatment/